CLINICAL TRIAL: NCT01788540
Title: The Role of Intralipid in Natural Killer Cell Positive Cases With Recurrent Miscarriages Undergoing IVF/ICSI Cycles: a Double Blind Randomized Controlled Trial
Brief Title: Intralipid for Recurrent Miscarriage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Dina Mohamed Refaat Dakhly, M.D., Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12013
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Abortion, Spontaneous; Abortion, Habitual
Keywords: Recurrent miscarriage; Implantation failure; Intralipid; ICSI / IVF failure
MeSH Terms: conditions — Abortion, Spontaneous; Abortion, Habitual | interventions — soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intralipid (Experimental): IV infusion of intralipid 20% is administrated on the day of vaginal egg collection in a dose of 9 mg/ml total blood volume corresponding to intralipid 2 ml 20% diluted in 250 ml saline over 30-60 minutes.
  the intralipid infusion is then repeated within the one week of positive pregnancy test and every 2 weeks till end of first trimester
  Interventions: Drug: Intralipid
- Control (No Intervention): No intervention

INTERVENTIONS:
Drug: Intralipid — IV infusion of intralipid 20% is administrated on the day of vaginal egg collection in a dose of 9 mg/ml total blood volume corresponding to intralipid 2 ml 20% diluted in 250 ml saline over 30-60 minutes.the intralipid infusion is then repeated within the 1st week of positive pregnancy test and every 2 weeks till end of first trimester
  Other Names: intralipid 20%
  Arms: Intralipid

SUMMARY:
Intralipid infusion can improve the outcome in NK cells positive females with history of recurrent miscarriages undergoing IVF/ICSI cycles.

ELIGIBILITY:
Inclusion Criteria:

* Couples with unexplained secondary infertility
* Three or more prior consecutive clinical miscarriages after either spontaneous pregnancy or after IVF/ICSI.
* Elevated natural killer (NK) cells CD16, CD56 and cells with both CD16/CD56 >12%.

Exclusion Criteria:

* Age above forty years old.
* Antiphospholipid syndrome (lupus anticoagulant and/or anticardiolipin antibodies [IgG or IgM]); other recognised thrombophilic conditions (testing according to usual clinic practice).
* Intrauterine abnormalities (as assessed by ultrasound, hysterosonography, hysterosalpingogram, or hysteroscopy).
* Abnormal parental karyotype.
* Other identifiable causes of recurrent miscarriages (tests initiated only if clinically indicated) e.g., diabetes, thyroid disease and systemic lupus erythematosus (SLE).
* Disturbances of normal fat metabolism such as pathologic hyperlipemia
* Allergic to it; or to eggs, soybean oil, or safflower oil.
* Severe liver disease, kidney disease, lung disease, anemia, blood clotting disorder.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-02; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
chemical pregnancy rate | 10 months
  Positive pregnancy test in blood as measured by quantitative B- hCG level

SECONDARY OUTCOMES:
clinical pregnancy rate, | 10 months
  Confirmed pregnancy at 7 weeks by ultrasound visualization of gestational sac and positive fetal pulsations

OTHER OUTCOMES:
ongoing pregnancy rate | 10 months
  clinical pregnancy continue after 12 weeks gestational age
abortion rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dina M Dakhly, M.D., Principal Investigator — Cairo University
Locations (1):
- Kasr el ainy hospital, Cairo, Egypt

REFERENCES:
- [Derived] Dakhly DM, Bayoumi YA, Sharkawy M, Gad Allah SH, Hassan MA, Gouda HM, Hashem AT, Hatem DL, Ahmed MF, El-Khayat W. Intralipid supplementation in women with recurrent spontaneous abortion and elevated levels of natural killer cells. Int J Gynaecol Obstet. 2016 Dec;135(3):324-327. doi: 10.1016/j.ijgo.2016.06.026. Epub 2016 Aug 30. PMID 27614789